CLINICAL TRIAL: NCT00003501
Title: Phase II Study of Antineoplaston A10 and AS2-1 in Patients With Non-Hodgkin's Lymphoma, High Grade
Brief Title: Antineoplaston Therapy in Treating Patients With High-Grade Stage II - Stage IV Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066541; BC-LY-08 (Other: Burzynski Research Institute)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Non-hodgkins Lymphoma
Keywords: Refractory Non-Hodgkin's Lymphoma; Recurrent Non-Hodgkin's Lymphoma; High-Grade Stage II - IV Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Antineoplaston therapy (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Patients with Refractory or Recurrent High-Grade Stage II - IV Non-Hodgkin's Lymphoma will receive Antineoplaston therapy (Atengenal + Astugenal).
  The daily doses of A10 and AS2-1 are divided into six infusions, which are given at 4-hourly intervals. Each infusion starts with infusion of A10 and is immediately followed by infusion of AS2-1.
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)

SUMMARY:
Current therapies for Refractory or Recurrent High-Grade Stage II - IV Non-Hodgkin's Lymphoma provide very limited benefit to the patient. The anti-cancer properties of Antineoplaston therapy suggest that it may prove beneficial in the treatment of Refractory or Recurrent High-Grade Stage II - IV Non-Hodgkin's Lymphoma.

PURPOSE: This study is being performed to determine the effects (good and bad) that Antineoplaston therapy has on patients with Refractory or Recurrent High-Grade Stage II - IV Non-Hodgkin's Lymphoma.

DETAILED DESCRIPTION:
Refractory or Recurrent High-Grade Stage II - IV Non-Hodgkin's Lymphoma patients receive gradually escalating doses of intravenous Antineoplaston therapy (Atengenal + Astugenal) until the maximum tolerated dose is reached. Treatment continues up to12 months in the absence of disease progression or unacceptable toxicity.

OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in patients with Refractory or Recurrent High-Grade Stage II - IV Non-Hodgkin's Lymphoma, as measured by an objective response to therapy (complete response, partial response or stable disease).
* To determine the safety and tolerance of Antineoplaston therapy in patients with Refractory or Recurrent High-Grade Stage II - IV Non-Hodgkin's Lymphoma.
* To determine objective response, tumor size is measured utilizing physical examination, radiologic studies, and bone marrow biopsies as necessary, performed every 8 weeks for the first two years, every 3 months for the third and fourth years, every 6 months for the 5th and sixth years, and annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven stage II, III, or IV high-grade non-Hodgkin's lymphoma that has not responded to, or has relapsed after a standard primary chemotherapy regimen plus at least 1 standard second-line salvage chemotherapy regimen NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adoptedby PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* WBC greater than 2000/mm^3
* Platelet count greater than 50,000/mm^3

Hepatic:

* Bilirubin no greater than 2.5 mg/dL

Renal:

* Creatinine no greater than 2.5 mg/dL
* No history of renal conditions that contraindicate high dosages of sodium

Cardiovascular:

* No uncontrolled hypertension
* No history of congestive heart failure
* No history of cardiovascular conditions that contraindicate high dosages of sodium

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study participation
* No active infection requiring treatment

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered
* No concurrent immunomodulatory agent (e.g., interferon or interleukin-2)

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered
* No concurrent antineoplastic agent

Endocrine therapy:

* At least 4 weeks since prior dexamethasone, prednisone, or other corticosteroids
* No concurrent corticosteroid

Radiotherapy:

* At least 8 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Other:

* No prior antineoplaston therapy
* No concurrent antibiotics, antifungals, or antivirals

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 1996-04-10 (Actual); Primary Completion 2003-07-02 (Actual); Study Completion 2003-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States